CLINICAL TRIAL: NCT04089722
Title: Efficacy and Safety of Deoxycholic Acid Injections for Removal of Adipose Tissue in the Anterior and Posterior Aspect of the Axilla "Bra Strap Fat"
Brief Title: Efficacy and Safety of Deoxycholic Acid Injections for Removal of Adipose Tissue in the "Bra Strap Fat" Region
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Juva Skin & Laser Center (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, Bruce E. Katz, Medical Director, Juva Skin & Laser Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 60E56
Record Dates: First submitted 2019-09-11; First posted 2019-09-13 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Brassiere Strap Fat (BSF); Bra Strap Fat (BSF)
MeSH Terms: interventions — Deoxycholic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Open-Label: Deoxycholic Acid Injections (Other): Deoxycholic Acid Injections (dose strength: 2 mg/cm2) via subcutaneous injections into posterior and/or anterior axillary roll adiposity. Patients will receive 10 mL or less (≤100 mg) of study drug per treatment administered in 0.2-mL injections with a 30-gauge, 0.5-in needle attached to a 1-mL syringe at 1.0-cm spacing using a customized grid. Up to 6 treatments (30 ± 7 days apart) will be permitted, but fewer can be allowed because of efficacy (insufficient BSF to inject, patient satisfaction with treatment) or safety/tolerability concerns.
  Interventions: Drug: Deoxycholic Acid

INTERVENTIONS:
Drug: Deoxycholic Acid — The active ingredient in KYBELLA® is synthetic deoxycholic acid. Deoxycholic acid is a naturally occurring molecule in the body that aids in the breakdown and absorption of dietary fat.
  Other Names: Kybella

SUMMARY:
This study evaluates the safety and efficacy of deoxycholic acid injections to dissolve adipose tissue in the anterior and posterior aspect of the axilla or the so called "brassiere strap fat" (BSF). Adult females aged 18-65 dissatisfied with their moderate or severe BSF will receive deoxycholic acid (dose strength: 2 mg/cm2) via subcutaneous injections into posterior and/or anterior axillary roll adiposity .

DETAILED DESCRIPTION:
The efficacy and safety of deoxycholic acid injections to dissolve adipose tissue in the submental area have been extensively evaluated. Deoxycholic acid injections have also been used successfully off-label to dissolve adipose tissues in other body areas. Our clinical experience in addition to a few case reports have shown the effectiveness and safety of deoxycholic acid injections to dissolve the adipose tissue in the anterior and posterior aspect of the axilla or the so called "brassiere strap fat" (BSF).

This is a single-center, prospective, single-arm, single-blind trial study.

This study is expected to benefit the existing literature by potentially adding a new non-invasive injectable treatment to a condition of excessive adipose tissue in the anterior and posterior aspect of the axilla that until now could only be treated with invasive surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult female age 18-65
* Subject satisfaction rating score of 0 or 1
* Clinician reported BSF rating score of 2, 3 or 4
* Patient reported BSF rating score of 2, 3 or 4
* Able to follow study instructions and likely to complete all required visits, as assessed by the Investigator.
* Willing to withhold additional aesthetic therapies to the proposed treatment area.
* Negative urine pregnancy test
* Willing to use acceptable methods of contraception throughout the study
* Sign an IRB-approved Informed Consent Form prior to any study-related procedures being performed.

Exclusion Criteria:

* History of any intervention to treat BSF (eg, liposuction, surgery, lipolytic agents)
* History of trauma associated with the axillary or upper back area
* Severe Skin Laxity Grade or other anatomical feature as assessed within 28 d before randomization, for which reduction in BSF may, in the judgment of the investigator, result in an aesthetically unacceptable outcome
* Evidence of any cause of enlargement in the upper back/ axillary roll (eg, tumors, lipomas) other than localized BSF
* BMI greater than 35 kg/m2
* A result on coagulation tests (prothrombin time, partial thromboplastin time) obtained within 28 d before randomization indicating the presence of any clinically significant bleeding disorder
* Any medical condition (eg, respiratory, cardiovascular, hepatic, neurologic disease, thyroid dysfunction) that would interfere with assessment of safety or efficacy or compromise the patient's ability to undergo study procedures or give informed consent
* History of sensitivity to any components of the study drug
* History of sensitivity to topical or local anesthetics (eg, lidocaine, benzocaine, procaine)
* Pregnancy
* Lactation
* Presence of infection at the injection sites

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 22 (Actual)
Dates: Start 2019-07-26 (Actual); Primary Completion 2020-06-11 (Actual); Study Completion 2020-10-22 (Actual)

PRIMARY OUTCOMES:
Reduction of Anterior/Posterior Axilla Fat | 6 months
  Composite improvements of 1 or more grades in BSF observed on both the Clinician- and Patient-Reported BSF Rating Scales

CONTACTS AND LOCATIONS:
Overall Officials: Bruce E Katz, MD, Principal Investigator — Juva Skin & Laser Center
Locations (1):
- JUVA Skin & Laser Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No